CLINICAL TRIAL: NCT00586508
Title: A Phase II Trial of Enzastaurin in Combination With Bevacizumab in Adults With Recurrent Malignant Gliomas
Brief Title: Trial of Enzastaurin and Bevacizumab in Participants With Recurrent Malignant Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11394; H6Q-MC-S033 (Other: Eli Lilly and Company); NCT00559923 (obsolete NCT alias)
Record Dates: First submitted 2007-12-07; First posted 2008-01-04 (Estimated); Results first posted 2020-09-24 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — enzastaurin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enzastaurin + Bevacizumab (Experimental)
  Interventions: Drug: enzastaurin; Drug: bevacizumab; Drug: Enzyme-inducing antiepileptic drugs (EIAED); Drug: Non-enzyme inducing antiepileptic drugs (NEIAED)

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) loading dose then 500 or 875 mg, orally, daily, 4-week cycles with participants evaluated after each cycle. The dose difference is for participants who are on enzyme-inducing antiepileptic drugs (EIAED) versus non-enzyme inducing antiepileptic drugs (NEIAED).
  Other Names: LY317615
Drug: bevacizumab — 10 milligrams per kilogram (mg/kg), intravenously (IV), every 2 weeks, participants are evaluated after each cycle (4-week cycles).
Drug: Enzyme-inducing antiepileptic drugs (EIAED) — Administered orally
Drug: Non-enzyme inducing antiepileptic drugs (NEIAED) — Administered orally

SUMMARY:
The purpose of this study is to evaluate both enzastaurin and bevacizumab in the treatment of recurrent malignant gliomas.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be at least 18 years old
* Participant must have been diagnosed with a recurrent brain tumor by magnetic resonance imaging (MRI) scan
* Participant must be willing to practice adequate contraception
* Participant must be able to swallow the enzastaurin tablets whole and receive bevacizumab intravenously
* Participant must agree to use the study drug only as instructed by your study doctor and staff.

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Participants who have significant heart, liver, kidney, or psychiatric disease
* Participants who have an active infection
* Participants who have any recent bleeding in the brain
* Participants who are taking any anti-coagulation or anti-platelet medication [including aspirin, non-steroidal anti-inflammatories, Cyclooxygenase-2 (COX-2) inhibitors]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bethesda, Maryland, United States

REFERENCES:
- [Derived] Odia Y, Iwamoto FM, Moustakas A, Fraum TJ, Salgado CA, Li A, Kreisl TN, Sul J, Butman JA, Fine HA. A phase II trial of enzastaurin (LY317615) in combination with bevacizumab in adults with recurrent malignant gliomas. J Neurooncol. 2016 Mar;127(1):127-35. doi: 10.1007/s11060-015-2020-x. Epub 2015 Dec 7. PMID 26643807
- [Derived] Odia Y, Shih JH, Kreisl TN, Fine HA. Bevacizumab-related toxicities in the National Cancer Institute malignant glioma trial cohort. J Neurooncol. 2014 Nov;120(2):431-40. doi: 10.1007/s11060-014-1571-6. Epub 2014 Aug 7. PMID 25098701
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The reasons for discontinuation listed in the participant flow are the reasons the participants discontinued treatment.
Groups:
- Enzastaurin + Bevacizumab (NEIAED): Enzastaurin: 1125 milligrams (mg) loading dose on Day 1, followed by 500 mg, orally, daily, for participants who are on non-enzyme inducing antiepileptic drugs (NEIAED) for 4 weeks. Participants were evaluated after each cycle (4-week cycles).
  Bevacizumab: 10 milligrams per kilogram (mg/kg), intravenously (IV), every 2 weeks. Participants were evaluated after each cycle (4-week cycles).
  Cycles repeated until there was evidence of progressive disease (PD), significant toxicity, withdrawal of consent, or other discontinuation criteria were met.
- Enzastaurin + Bevacizumab (EIAED): Enzastaurin: 1125 mg loading dose on Day 1, followed by 875 mg, orally, daily, for participants who are on enzyme inducing antiepileptic drugs (EIAED) for 4 weeks. Participants were evaluated after each cycle (4-week cycles).
  Bevacizumab: 10 mg/kg, IV, every 2 weeks. Participants were evaluated after each cycle (4-week cycles).
  Cycles repeated until there was evidence of PD, significant toxicity, withdrawal of consent, or other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Started | 68 | 13
Received at Least 1 Dose of Study Drug | 68 | 13
Completed | 0 | 0
Not Completed | 68 | 13
Not completed — Progressive disease | 52 | 8
Not completed — Death | 0 | 1
Not completed — Adverse Event | 12 | 4
Not completed — Withdrawal by Subject | 4 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- Enzastaurin + Bevacizumab (NEIAED): Enzastaurin: 1125 mg loading dose on Day 1, followed by 500 mg, orally, daily, for participants who are on NEIAED for 4 weeks. Participants were evaluated after each cycle (4-week cycles).
  Bevacizumab: 10 mg/kg, IV, every 2 weeks. Participants were evaluated after each cycle (4-week cycles).
  Cycles repeated until there was evidence of PD, significant toxicity, withdrawal of consent, or other discontinuation criteria were met.
- Enzastaurin + Bevacizumab (EIAED): Enzastaurin: 1125 mg loading dose on Day 1, followed by 875 mg, orally, daily, for participants who are on EIAED for 4 weeks. Participants were evaluated after each cycle (4-week cycles).
  Bevacizumab: 10 mg/kg, IV, every 2 weeks. Participants were evaluated after each cycle (4-week cycles).
  Cycles repeated until there was evidence of PD, significant toxicity, withdrawal of consent, or other discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED) | Total
Number analyzed (Participants) | 68 | 13 | 81
Age, Continuous [Median (Full Range); unit: years] | 50 (11.59) [25.40 to 72.70] | 44 (11.97) [26.50 to 66.10] | 49 (11.61) [25.40 to 72.70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 4 | 26
  Male | 46 | 9 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 68 | 13 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 0 | 6
  White | 58 | 13 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 13 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival at 6 Months (PFS-6)
Description: Data presented are the percentage of participants without progressive disease (PD) or death from any cause 6 months after registration. PD was a 25% increase in the sum of products of all measurable lesions (or 2 largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) or clear worsening of any evaluable disease, or appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer).
Time Frame: Registration to 6 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 68 | 13
percentage of participants | 31 [21 to 42] | 15 [2 to 39]

2. Primary Outcome: Time to Progressive Disease (PD)
Description: Defined as the time from registration to PD, death or date of last contact. PD was a 25% increase in the sum of products of all measurable lesions (or 2 largest lesions if too numerous) over the smallest sum observed (over baseline if no decrease) or clear worsening of any evaluable disease, or appearance of any new lesion/site, or failure to return for evaluation due to death or deteriorating condition (unless clearly unrelated to this cancer). Participants who had no PD or death at the time of the data inclusion cutoff, time to PD was censored at their last tumor assessment prior to the cutoff date.
Time Frame: Registration to PD, death or date of last contact up to 66.56 months
Population: All enrolled participants who received at least 1 dose of study drug. The number of participants censored are 7 for Enzastaurin + Bevacizumab NEIAED) group and 0 for Enzastaurin + Bevacizumab (EIAED) group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 68 | 13
months | 2.76 [2.00 to 4.37] | 1.84 [0.92 to 2.69]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall response is confirmed complete response (CR) + partial response (PR). CR is complete disappearance of all measurable and evaluable disease, no new lesions, and no evidence of non-evaluable disease. PR is ≥50% decrease compared to baseline in the sum of products of perpendicular diameters of all measurable lesions (or the 2 largest lesions), no progression of evaluable disease and no new lesions. ORR is calculated as (total number of participants with CR or PR from the start of registration until disease progression) / (the total number of participants treated)*100.
Time Frame: Registration to date of objective PD or death up to 66.56 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 68 | 13
percentage of participants | 5.9 [1.6 to 14.4] | 0 [NA to NA] — Zero participants had response; therefore 95% confidence interval was not calculated.

4. Secondary Outcome: To Evaluate Tumor Markers and Genes
Time Frame: Baseline and every cycle (4-week cycles)
Population: Data were not collected for any participant due to low samples.
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) Subscales
Description: HRQoL was assessed with the Functional Assessment of Cancer Therapy - Brain (FACT-Br) version 4. The instrument consists of 50 items with a 5-point rating scale for each item, where 0 = "not at all" and 4 = "very much." Physical well-being, social/family well-being and functional well-being subscales consist of 7 items each with scores ranging from 0-28. The emotional well-being subscale consists of 6 items with a score ranging from 0-24. The brain cancer-specific subscale consists of 23 items with a score ranging from 0-92. Higher scores in each subscale represent better QoL. Changes from baseline in the 4 core subscales are presented.
Time Frame: Baseline, Cycles 1-12 (4-week cycles)
Population: All enrolled participants who received at least 1 dose of study drug and had HRQoL assessed at baseline and in the end of Cycles 1-12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 68 | 13
units on a scale
  Physical Well-Being Cycle 1: number analyzed (Participants) | 25 | 4
  Physical Well-Being Cycle 1 | 1.4 (3.27) | 2.5 (4.04)
  Physical Well-Being Cycle 2: number analyzed (Participants) | 20 | 3
  Physical Well-Being Cycle 2 | 1.2 (3.15) | 2.0 (4.36)
  Physical Well-Being Cycle 3: number analyzed (Participants) | 16 | 2
  Physical Well-Being Cycle 3 | 2.3 (4.60) | -0.5 (0.71)
  Physical Well-Being Cycle 4: number analyzed (Participants) | 12 | 2
  Physical Well-Being Cycle 4 | 1.8 (3.49) | -3.0 (2.83)
  Physical Well-Being Cycle 5: number analyzed (Participants) | 9 | 2
  Physical Well-Being Cycle 5 | 1.0 (1.87) | 0.5 (0.71)
  Physical Well-Being Cycle 6: number analyzed (Participants) | 7 | 2
  Physical Well-Being Cycle 6 | -0.1 (3.02) | -1.0 (1.41)
  Physical Well-Being Cycle 7: number analyzed (Participants) | 5 | 1
  Physical Well-Being Cycle 7 | -1.4 (3.21) | 0.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Physical Well-Being Cycle 8: number analyzed (Participants) | 5 | 1
  Physical Well-Being Cycle 8 | 0.8 (1.92) | 0.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Physical Well-Being Cycle 9: number analyzed (Participants) | 5 | 0
  Physical Well-Being Cycle 9 | 0.2 (3.63) |
  Physical Well-Being Cycle 10: number analyzed (Participants) | 5 | 0
  Physical Well-Being Cycle 10 | 0.6 (4.67) |
  Physical Well-Being Cycle 11: number analyzed (Participants) | 5 | 0
  Physical Well-Being Cycle 11 | 0.2 (3.03) |
  Physical Well-Being Cycle 12: number analyzed (Participants) | 4 | 0
  Physical Well-Being Cycle 12 | -0.5 (2.08) |
  Social/Family Well-Being Cycle 1: number analyzed (Participants) | 25 | 4
  Social/Family Well-Being Cycle 1 | -0.2 (2.02) | 0.0 (0.82)
  Social/Family Well-Being Cycle 2: number analyzed (Participants) | 20 | 3
  Social/Family Well-Being Cycle 2 | 0.1 (2.13) | 0.3 (1.53)
  Social/Family Well-Being Cycle 3: number analyzed (Participants) | 16 | 2
  Social/Family Well-Being Cycle 3 | -0.1 (2.47) | 0.5 (0.71)
  Social/Family Well-Being Cycle 4: number analyzed (Participants) | 12 | 2
  Social/Family Well-Being Cycle 4 | -0.1 (2.50) | 1.0 (5.66)
  Social/Family Well-Being Cycle 5: number analyzed (Participants) | 9 | 2
  Social/Family Well-Being Cycle 5 | 0.2 (2.59) | -1.5 (2.12)
  Social/Family Well-Being Cycle 6: number analyzed (Participants) | 7 | 2
  Social/Family Well-Being Cycle 6 | 0.0 (1.91) | -1.0 (2.83)
  Social/Family Well-Being Cycle 7: number analyzed (Participants) | 5 | 1
  Social/Family Well-Being Cycle 7 | 0.0 (2.55) | -3.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Social/Family Well-Being Cycle 8: number analyzed (Participants) | 5 | 1
  Social/Family Well-Being Cycle 8 | -1.2 (1.30) | -3.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Social/Family Well-Being Cycle 9: number analyzed (Participants) | 5 | 0
  Social/Family Well-Being Cycle 9 | 1.6 (4.04) |
  Social/Family Well-Being Cycle 10: number analyzed (Participants) | 5 | 0
  Social/Family Well-Being Cycle 10 | 0.2 (1.30) |
  Social/Family Well-Being Cycle 11: number analyzed (Participants) | 5 | 0
  Social/Family Well-Being Cycle 11 | 1.2 (2.28) |
  Social/Family Well-Being Cycle 12: number analyzed (Participants) | 4 | 0
  Social/Family Well-Being Cycle 12 | 2.5 (3.11) |
  Emotional Well-Being Cycle 1: number analyzed (Participants) | 25 | 4
  Emotional Well-Being Cycle 1 | 0.1 (5.44) | -1.8 (2.50)
  Emotional Well-Being Cycle 2: number analyzed (Participants) | 20 | 3
  Emotional Well-Being Cycle 2 | -1.5 (2.86) | -4.0 (2.65)
  Emotional Well-Being Cycle 3: number analyzed (Participants) | 16 | 2
  Emotional Well-Being Cycle 3 | -0.8 (3.86) | -4.5 (0.71)
  Emotional Well-Being Cycle 4: number analyzed (Participants) | 12 | 2
  Emotional Well-Being Cycle 4 | -1.3 (2.49) | -3.5 (0.71)
  Emotional Well-Being Cycle 5: number analyzed (Participants) | 9 | 2
  Emotional Well-Being Cycle 5 | -1.3 (3.43) | -1.0 (4.24)
  Emotional Well-Being Cycle 6: number analyzed (Participants) | 7 | 2
  Emotional Well-Being Cycle 6 | -1.9 (3.85) | 0.0 (5.66)
  Emotional Well-Being Cycle 7: number analyzed (Participants) | 5 | 1
  Emotional Well-Being Cycle 7 | -4.2 (3.56) | -4.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Emotional Well-Being Cycle 8: number analyzed (Participants) | 5 | 1
  Emotional Well-Being Cycle 8 | -2.4 (2.51) | -2.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Emotional Well-Being Cycle 9: number analyzed (Participants) | 5 | 0
  Emotional Well-Being Cycle 9 | -1.8 (1.79) |
  Emotional Well-Being Cycle 10: number analyzed (Participants) | 5 | 0
  Emotional Well-Being Cycle 10 | -0.6 (5.41) |
  Emotional Well-Being Cycle 11: number analyzed (Participants) | 5 | 0
  Emotional Well-Being Cycle 11 | -2.0 (2.45) |
  Emotional Well-Being Cycle 12: number analyzed (Participants) | 4 | 0
  Emotional Well-Being Cycle 12 | -1.3 (3.59) |
  Functional Well-Being Cycle 1: number analyzed (Participants) | 25 | 4
  Functional Well-Being Cycle 1 | 0.7 (6.57) | 3.0 (4.76)
  Functional Well-Being Cycle 2: number analyzed (Participants) | 20 | 3
  Functional Well-Being Cycle 2 | 0.3 (5.58) | 1.0 (4.36)
  Functional Well-Being Cycle 3: number analyzed (Participants) | 16 | 2
  Functional Well-Being Cycle 3 | 0.1 (5.41) | 1.0 (1.41)
  Functional Well-Being Cycle 4: number analyzed (Participants) | 12 | 2
  Functional Well-Being Cycle 4 | -0.3 (2.19) | 3.0 (1.41)
  Functional Well-Being Cycle 5: number analyzed (Participants) | 9 | 2
  Functional Well-Being Cycle 5 | -1.4 (3.64) | 0.5 (2.12)
  Functional Well-Being Cycle 6: number analyzed (Participants) | 7 | 2
  Functional Well-Being Cycle 6 | -2.9 (6.18) | -2.5 (6.36)
  Functional Well-Being Cycle 7: number analyzed (Participants) | 5 | 1
  Functional Well-Being Cycle 7 | -2.6 (5.86) | 2.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Functional Well-Being Cycle 8: number analyzed (Participants) | 5 | 1
  Functional Well-Being Cycle 8 | -3.8 (4.71) | 3.0 (NA) — 1 participant was analyzed; therefore actual value was presented and standard deviation was not calculated.
  Functional Well-Being Cycle 9: number analyzed (Participants) | 5 | 0
  Functional Well-Being Cycle 9 | -1.8 (3.56) |
  Functional Well-Being Cycle 10: number analyzed (Participants) | 5 | 0
  Functional Well-Being Cycle 10 | -3.6 (5.22) |
  Functional Well-Being Cycle 11: number analyzed (Participants) | 5 | 0
  Functional Well-Being Cycle 11 | -1.8 (4.44) |
  Functional Well-Being Cycle 12: number analyzed (Participants) | 4 | 0
  Functional Well-Being Cycle 12 | -3.0 (4.55) |
Statistical Analysis 1: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.3375, ANCOVA — P-value is for Physical Well-Being Cycle 1; P-value of treatment effect from an Analysis of Covariance (ANCOVA) for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 2: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.516, ANCOVA — P-value is for Physical Well-Being Cycle 2; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 3: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.786, ANCOVA — P-value is for Physical Well-Being Cycle 3; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 4: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.1496, ANCOVA — P-value is for Physical Well-Being Cycle 4; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 5: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8428, ANCOVA — P-value is for Physical Well-Being Cycle 5; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 6: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7345, ANCOVA — P-value is for Physical Well-Being Cycle 6; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 7: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8928, ANCOVA — P-value is for Physical Well-Being Cycle 7; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 8: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7343, ANCOVA — P-value is for Physical Well-Being Cycle 8; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 9: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8798, ANCOVA — P-value is for Social/Family Well-Being Cycle 1; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 10: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.6837, ANCOVA — P-value is for Social/Family Well-Being Cycle 2; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 11: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7226, ANCOVA — P-value is for Social/Family Well-Being Cycle 3; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 12: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.641, ANCOVA — P-value is for Social/Family Well-Being Cycle 4; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 13: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.478, ANCOVA — P-value is for Social/Family Well-Being Cycle 5; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 14: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.9367, ANCOVA — P-value is for Social/Family Well-Being Cycle 6; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 15: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.5108, ANCOVA — P-value is for Social/Family Well-Being Cycle 7; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 16: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8976, ANCOVA — P-value is for Social/Family Well-Being Cycle 8; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 17: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8193, ANCOVA — P-value is for Emotional Well-Being Cycle 1; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 18: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.1695, ANCOVA — P-value is for Emotional Well-Being Cycle 2; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 19: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.4021, ANCOVA — P-value is for Emotional Well-Being Cycle 3; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 20: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.3603, ANCOVA — P-value is for Emotional Well-Being Cycle 4; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 21: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.5169, ANCOVA — P-value is for Emotional Well-Being Cycle 5; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 22: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.1642, ANCOVA — P-value is for Emotional Well-Being Cycle 6; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 23: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.6354, ANCOVA — P-value is for Emotional Well-Being Cycle 7; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 24: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.3517, ANCOVA — P-value is for Emotional Well-Being Cycle 8; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 25: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7605, ANCOVA — P-value is for Functional Well-Being Cycle 1; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 26: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.3747, ANCOVA — P-value is for Functional Well-Being Cycle 2; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 27: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.8379, ANCOVA — P-value is for Functional Well-Being Cycle 3; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 28: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.1179, ANCOVA — P-value is for Functional Well-Being Cycle 4; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 29: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7412, ANCOVA — P-value is for Functional Well-Being Cycle 5; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 30: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.3773, ANCOVA — P-value is for Functional Well-Being Cycle 6; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 31: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.7402, ANCOVA — P-value is for Functional Well-Being Cycle 7; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value
Statistical Analysis 32: Comparison: Enzastaurin + Bevacizumab (NEIAED) vs Enzastaurin + Bevacizumab (EIAED); Test type: Superiority or Other; p = 0.2671, ANCOVA — P-value is for Functional Well-Being Cycle 8; P-value of treatment effect from an ANCOVA for change from baseline. Covariates include: treatment and baseline value

6. Primary Outcome: Number of Participants With Adverse Events (AEs) or Deaths (Safety)
Description: Data presented are the number of participants who experienced serious adverse events (SAEs), other non-serious AEs and deaths during the study including the 30-day follow-up. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Event module.
Time Frame: Registration to study completion up to 67.56 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Number analyzed (Participants) | 68 | 13
Participants
  SAEs | 24 | 4
  AEs | 68 | 13
  Deaths | 5 | 1

ADVERSE EVENTS:
Arm/Group | Enzastaurin + Bevacizumab (NEIAED) | Enzastaurin + Bevacizumab (EIAED)
Serious Adverse Events (participants affected / at risk) | 24/68 | 4/13
Other Adverse Events (participants affected / at risk) | 68/68 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin + Bevacizumab (NEIAED) (N=68) | Enzastaurin + Bevacizumab (EIAED) (N=13)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Death (General disorders) | 2 (2) | 0 (0)
Disease progression (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 0 (0) | 1 (1)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0)
Blood sodium increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 7 (7) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin + Bevacizumab (NEIAED) (N=68) | Enzastaurin + Bevacizumab (EIAED) (N=13)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Cushingoid (Endocrine disorders) | 4 (4) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 14 (14) | 2 (2)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 0 (0)
Fatigue (General disorders) | 25 (25) | 4 (4)
Medical device complication (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 5 (5) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 4 (4) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 18 (18) | 2 (2)
Blood albumin decreased (Investigations) | 7 (7) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 8 (8) | 1 (1)
Blood bilirubin increased (Investigations) | 7 (7) | 1 (1)
Blood creatinine increased (Investigations) | 5 (5) | 0 (0)
Blood glucose increased (Investigations) | 4 (4) | 0 (0)
Blood magnesium decreased (Investigations) | 4 (4) | 0 (0)
Blood magnesium increased (Investigations) | 23 (23) | 2 (2)
Blood phosphorus decreased (Investigations) | 18 (18) | 2 (2)
Blood potassium increased (Investigations) | 13 (13) | 4 (4)
Blood sodium decreased (Investigations) | 15 (15) | 2 (2)
Blood sodium increased (Investigations) | 9 (9) | 2 (2)
Blood uric acid increased (Investigations) | 7 (7) | 0 (0)
Haemoglobin decreased (Investigations) | 15 (15) | 3 (3)
Laboratory test abnormal (Investigations) | 9 (9) | 2 (2)
Lymphocyte count decreased (Investigations) | 37 (37) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (6) | 2 (2)
Platelet count decreased (Investigations) | 25 (25) | 3 (3)
Protein urine present (Investigations) | 15 (15) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 8 (8) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 13 (16) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 13 (13) | 1 (1)
Headache (Nervous system disorders) | 9 (9) | 1 (1)
Memory impairment (Nervous system disorders) | 4 (4) | 0 (0)
Nervous system disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1)
Speech disorder (Nervous system disorders) | 9 (9) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 5 (5) | 1 (1)
Chromaturia (Renal and urinary disorders) | 11 (11) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 5 (5) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 2/22 (2) | 0/4 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0/22 (0) | 1/4 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/22 (0) | 1/4 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 (10) | 1 (1)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 8 (8) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hypertension (Vascular disorders) | 14 (14) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days